CLINICAL TRIAL: NCT06705452
Title: 4D-MRI Morphological Study of Local Growth in Cerebral Aneurysms
Brief Title: MRI Analysis in the Growth of Cerebral Aneurysms
Acronym: EPICAVC
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PO24101
Record Dates: First submitted 2024-11-22; First posted 2024-11-26 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-11

CONDITIONS: Unruptured Intracranial Aneurysm
Keywords: Aneurysm Growth; Unruptured Intracranial aneurysm; Cerebral Aneurysm; Vascular Diseases; Intracranial Arterial Diseases; Intracranial Aneurysm
MeSH Terms: conditions — Intracranial Aneurysm; Vascular Diseases; Intracranial Arterial Diseases

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with unruptured and untreated aneurysms (Experimental): Patients in radiology for the first diagnostic evaluation or the follow-up of unruptured and untreated aneurysms.
  Interventions: Other: Additional 4D Flow MRI or additional 4D Flow sequence

INTERVENTIONS:
Other: Additional 4D Flow MRI or additional 4D Flow sequence — Additional 4D Flow MRI or additional 4D Flow sequence

SUMMARY:
An intracranial aneurysm is defined as a localized dilatation of the cerebral arteries, which can potentially lead to rupture and subsequent hemorrhagic stroke. The mechanisms by which aneurysms develop and grow remain unknown. The objective of this project is to utilize MRI, a routine non-invasive examination for detecting and following up aneurysms, to identify visually and quantitatively an aneurysm growth and relevant biomarkers that can predict the risk of aneurysm development.

DETAILED DESCRIPTION:
An intracranial aneurysm is defined as a malformation of the cerebral arteries, which is characterized by a focal dilatation of the arterial wall.

The prevalence of intracranial aneurysms in the general population is estimated to be between 3% and 6%, as reported in the literature. Although the rupture rate is relatively low, at approximately 1-2% per year per aneurysm, this risk is increased if the aneurysm is growing. The morbi-mortality rates associated with meningeal or subarachnoid hemorrhage are high, with an estimated 60% mortality rate within three months and 30% of patients remaining permanently disabled. It is therefore imperative to monitor the evolution of aneurysms in order to assess the risk of complications and guide therapeutic decisions.

The mechanism(s) of aneurysm formation and growth remain unknown. Aneurysms form in a zone of weakness in the artery wall as a result of hemodynamic variations.

Methods of risk stratification and therapeutic planning (endovascular treatment (coil) or surgical treatment (clip)) are currently based solely on empirical and statistical parameters such as the size or shape of the aneurysm, the patient's smoking habits or alcoholism.

The fundamental principle underlying the treatment of cerebral aneurysms with the objective of reducing the risk of long-term rupture is the exclusion of the aneurysm from the arterial circulation. This confirm the impact of hemodynamics on the risk of aneurysm rupture.

Although arteriography remains the gold standard for follow-up of aneurysms, it is an invasive and irradiative examination that is increasingly being replaced by a non-invasive routine exam, Magnetic Resonance Imaging (MRI).

Currently, there is no consensus regarding the indications for the treatment of unruptured intracranial aneurysms, which are generally asymptomatic. Successful outcome of the project would improve physical understanding of aneurysmal pathology, enabling the decision-making process regarding treatment to be adapted to the specific characteristics of the aneurysm in question. This would provide additional arguments for proposing or not proposing expensive endovascular treatment of aneurysms, which is often proposed as a first-line treatment.

ELIGIBILITY:
inclusion criteria:

* Patients with one or more unruptured intracranial aneurysms followed up at the participating center. Patients may have other ruptured and/or treated aneurysms
* Patient older than 18 years
* Patient consenting to participate to the study
* Patient enrolled in the national healthcare insurance program

exclusion criteria:

* Patients who have already received surgical or endovascular treatment for all their aneurysm(s), or who are due to receive such treatment in less than 2 months.
* Patients with only ruptured aneurysm(s)
* Patients with arteriovenous malformations (treated or untreated)
* Patients with a contraindication to MRI
* Patients with an allergy to one of the contrast agents (Iodixanol, Gadoteric acid)
* Pregnant or breast-feeding patients
* Patients protected by law.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 281 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2031-01-01 (Estimated); Study Completion 2032-01-01 (Estimated)

PRIMARY OUTCOMES:
Evolution of the shape of the aneurysm | At 3 years
  Millimetric quantification of the three-dimensional evolution of the shape of the aneurysm sac, calculated using a computer algorithm

CONTACTS AND LOCATIONS:
Locations (1):
- Damien JOLLY, Reims, France